CLINICAL TRIAL: NCT06518434
Title: A Phase 2a Study on the Anti-tumoral Effect of Cannabis Oil (THC 10% / CBD 5%) in Patients With Advanced Untreatable Hepatocellular Carcinoma
Brief Title: A Pilot Study on the Effect of Cannabis Oil in Untreatable Liver Cancer Patients
Acronym: CanHep
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten Nijkamp, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201800881
Record Dates: First submitted 2021-09-28; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma; Cannabis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Marijuana Abuse | interventions — Medical Marijuana; Dronabinol; Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabis oil (Experimental): Treatment with cannabis oil
  Interventions: Drug: Medical Cannabis

INTERVENTIONS:
Drug: Medical Cannabis — Medical cannabis oil three times daily
  Other Names: Cannabis oil containing 10% delta-9-tetrahydrocannabinol (THC) and 5% cannabidiol (CBD)

SUMMARY:
to study the anti-tumor effect of cannabis oil (THC10% / CBD5%) in untreatable HCC patients based on mRECIST and RECIST criteria

ELIGIBILITY:
Inclusion Criteria:

* Age =>18 yrs
* Histologically proven hepatocellular carcinoma
* Non-cirrhosis or Child Pugh A cirrhosis
* Hepatic encephalopathy grade 0 or 1
* Multidisciplinary treatment (MDT)-advised best supportive care for untreatable advanced HCC or patients unable to undergo or declining treatment for advanced HCC.
* Minimal life expectancy of 3 months
* Willing and able to attend follow-up examinations
* Willing to stop active traffic participation or controlling machinery during the study period if applicable
* Signed informed consent
* Language: Dutch or English

Exclusion Criteria:

* Child Pugh B or C cirrhosis
* Hepatic encephalopathy grade 2 or more
* Previous systemic treatment for HCC
* Mental conditions rendering the subject incapable to understand the nature, scope and consequences of the trial
* Use of medicinal cannabis for other purposes
* Contra-indications for medicinal cannabis oil:

  * Patients who have experienced a myocardial infarction or clinically significant cardiac dysfunction within the last 12 months or have had a cardiac disorder that, in the opinion of the investigator would have put the participant at risk of a clinically significant arrhythmia or myocardial infarction.
  * Patients with known psychotic disorders
  * Female patients who are pregnant or lactating
  * Patients (men or women) intending to start a family
  * Hypersensitivity to cannabinoids or any of the excipients of the cannabis oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Tumor size | 9 months
  Tumor size based on RECIST and mRECIST criteria

SECONDARY OUTCOMES:
Tumor size | 3 months
  Tumor size based on RECIST and mRECIST criteria
Tumor size | 6 months
  Tumor size based on RECIST and mRECIST criteria
Tumor markers | 3 months
  Alfa-foetoprotein (AFP) and des-gamma-carboxy-protrombine (DGCPT)
Tumor markers | 6 months
  Alfa-foetoprotein (AFP) and des-gamma-carboxy-protrombine (DGCPT)
Tumor markers | 9 months
  Alfa-foetoprotein (AFP) and des-gamma-carboxy-protrombine (DGCPT)
Quality of Life questionnaires | 3 months
  EORTC-QLQ30 and -HCC18
Quality of Life questionnaires | 6 months
  EORTC-QLQ30 and -HCC18
Quality of Life questionnaires | 9 months
  EORTC-QLQ30 and -HCC18

CONTACTS AND LOCATIONS:
Overall Officials: M W Nijkamp, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No